CLINICAL TRIAL: NCT03677375
Title: Hemodilution Validation of INVSENSOR00026
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP-19466
Record Dates: First submitted 2018-09-17; First posted 2018-09-19 (Actual); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-04

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Test Subject (Experimental): All subjects who are enrolled into the test group and participate in data collection receive the noninvasive INVSENSOR00026.
  Interventions: Device: INVSENSOR00026

INTERVENTIONS:
Device: INVSENSOR00026 — Noninvasive pulse oximeter sensor

SUMMARY:
In this study, the concentration of hemoglobin within the subject's blood will be reduced in a controlled manner by administering fluids intravenously. The accuracy of a noninvasive hemoglobin sensor will be assessed by comparison to hemoglobin measurements from a laboratory analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Subject weighs a minimum of 110 lbs and no more than 250 lbs unless subject is over 6 feet tall.
* Hemoglobin value is greater than or equal to 11 g/dL at time of screening
* Baseline heart rate ≥ 45 bpm and ≤ 85 bpm.
* CO value ≤ 2.0% FCOHb
* Subject has a physical status of ASA I or II (American Society of Anesthesiology Class I; Healthy subjects without any systemic disease at all. American Society of Anesthesiology Class II; subjects with mild systemic disease) as it applies to the systemic disease portion of the classification.
* Systolic Blood Pressure ≤ 140 mmHg and Diastolic Blood Pressure ≤ 90 mmHg.
* Subject is able to read and communicate in English and understands the study and risks involved.

Exclusion Criteria:

* Subject is pregnant
* Subject smokes (including e-cigarette use)
* Subject has a BMI > 35 and has been classified as morbidly obese or at an increased risk for participation by a medical professional.
* Subject has a history of fainting (vasovagal), blacking out or losing consciousness during or after a blood draw.
* Subject has open wounds, inflamed tattoos or piercings, or any visible healing wounds.
* Subject has known drug or alcohol abuse or uses recreational drugs.
* Subject has experienced a head injury with loss of consciousness within the last year.
* Subject has taken anticoagulant medication within the last 30 days.
* Subject has any chronic bleeding disorders (i.e. hemophilia).
* Subject has any history of a stroke, myocardial infarction, heart attack, or seizures.
* Subject has any cancer or history of cancer (not including skin cancer).
* Subject has a chronic neurological disease (i.e. multiple sclerosis, Huntington's disease).
* Subject has any cardiac dysrhythmias (i.e. atrial fibrillation) and has not received clearance from their physician.
* Subject has known neurological and/or psychiatric disorder (i.e. schizophrenia, bipolar disorder) that interferes with the subject's level of consciousness.
* Subject has Wolff-Parkinson-White Syndrome or Stokes-Adams Syndrome
* Subject has any medical condition which in the judgment of the investigator and/or medical staff, renders them ineligible for participation in this study (Discretion of investigator).
* Subject has taken opioid pain medication within 24 hours of start of study.
* Subject has any type of infectious disease (i.e. Hepatitis, HIV, Tuberculosis, Flu, Malaria, Measles, etc.).
* Subject is taking medications known to treat any type of infectious disease.
* Subject has either signs or history of peripheral ischemia or carpal tunnel.
* Subject has had invasive surgery within the past year- including but not limited to major dental surgery, gallbladder, heart, appendix, major fracture repairs (involving plates/ screws), jaw surgery, Urinary tract surgery, plastic surgery, major ENT surgery, joint replacement or gynecological surgeries, heart surgery or thoracic surgery.
* Subject has symptoms of congestion, head colds, flu, or other illnesses
* Subject has donated blood within the last 2 weeks.
* Subject is claustrophobic or has generalized anxiety disorder.
* Subject has been in severe car accident(s) or a similar type of accident(s) requiring hospitalization within the last 12 months.
* Subject has had a concussion within the last 12 months.
* Subject has chronic unresolved asthma, lung disease or respiratory disease.
* Subject is allergic to lidocaine, latex, adhesives, or plastic.
* Subject has heart conditions, insulin-dependent diabetes or uncontrolled hypertension.
* Subject has delivered vaginally, has had a pregnancy terminated, a miscarriage with hospitalization, or had a C-section within the last 6 months.
* Subject intends on participating in any heavy lifting, repetitive movement of their wrist (including riding a motorcycle) or exercise (working out, riding a bike, riding a skate board etc.), or any activity that will put additional stress on the wrist within 24 hours following a study that involves an arterial line.
* Discretion of investigator/study staff

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 173 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-02-04 (Actual); Study Completion 2019-02-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Masimo Corporation, Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol enrollment number includes screen failures and subjects that did not proceed due to time constraints
Period: Overall Study
Arm/Group | Test Subject
Started | 93
Completed | 81
Not Completed | 12
Not completed — Incomplete procedure | 8
Not completed — Adverse Event | 3
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Population: Subjects whose hemoglobin levels did not meet predefined study requirements were not included in the final data analysis.
Arm/Group | Test Subject
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 40
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian or Pacific Islander | 4
  Caucasian | 15
  Black or African American | 12
  Hispanic | 9

OUTCOME MEASURES:

1. Primary Outcome: Accuracy of Noninvasive Hemoglobin Sensor by Arms Calculation
Description: Accuracy will be determined by comparing the noninvasive hemoglobin measurement of the pulse oximeter to the hemoglobin value obtained from a blood sample and calculating the arithmetic root mean square (Arms) error value. In order to obtain the Arms value, the blood sample hemoglobin value is subtracted from the pulse oximeter hemoglobin value for a number of samples, the average of this difference is computed as the bias. The standard deviation of the differences is computed as the precision. The square root of the sum of the squares of bias and precision is computed as the Arms Error value.
Time Frame: 1-5 hours
Measure: Number; unit: g/dL
Arm/Group | Test Subject
Number analyzed (Participants) | 40
g/dL | 1.13

ADVERSE EVENTS:
Time Frame: 5 months
Arm/Group | Test Subject
All-Cause Mortality (participants affected / at risk) | 0/93
Serious Adverse Events (participants affected / at risk) | 0/93
Other Adverse Events (participants affected / at risk) | 8/93
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Subject (N=93)
Swelling due to IV catheter site infiltration (Injury, poisoning and procedural complications) | 2
Vasovagal episode during arterial line placement (Injury, poisoning and procedural complications) | 1
Numbness secondary to local anesthetic infiltration (Injury, poisoning and procedural complications) | 1
Bruising and swelling at arterial site (Injury, poisoning and procedural complications) | 2
Headache (Injury, poisoning and procedural complications) | 1
Discomfort (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/75/NCT03677375/Prot_SAP_000.pdf